CLINICAL TRIAL: NCT00892970
Title: The Effects of Azithromycin Ophthalmic Solution, 1% Versus Placebo in Subjects With Blepharitis During a Two-Week Treatment Period
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Mike Schiewe, Inspire
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 044-101; P08639
Record Dates: First submitted 2009-05-01; First posted 2009-05-05 (Estimated); Last update posted 2011-09-26 (Estimated); Status verified 2011-09

CONDITIONS: Blepharitis
MeSH Terms: conditions — Blepharitis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- 1 (Experimental)
  Interventions: Drug: Azithromycin ophthalmic solution, 1%
- 2 (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Azithromycin ophthalmic solution, 1% — One drop in each eye twice a day for the first two days; then one drop in each eye once a day for 12 days
  Arms: 1
Drug: Placebo — One drop in each eye twice a day for the first two days; then one drop in each eye once a day for 12 days
  Arms: 2

SUMMARY:
The objective of this study is to compare the safety and efficacy of azithromycin ophthalmic solution, 1% versus placebo over a two-week treatment period.

ELIGIBILITY:
Inclusion Criteria:

* Have best corrected visual acuity in both eyes of at least +0.7 or better
* If female, are non-pregnant or non-lactating
* Have a current diagnosis of blepharitis in one or both eyes

Exclusion Criteria:

* Have lid structural abnormalities
* Have suspected ocular fungal or viral infection
* Have practiced warm compress therapy within 14 days prior to Visit 2
* Unable to withhold the use of contact lenses during the treatment or follow-up periods
* Unable to withhold the use of ocular cosmetic products within 24 hours prior to study visits
* Have had penetrating intraocular surgery within 90 days prior to Visit 2
* Have had ocular surface surgery within the past year prior to Visit 2
* Have a serious medical condition which could confound study assessments

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 313 (Actual)
Dates: Start 2009-04; Primary Completion 2010-01 (Actual); Study Completion 2010-01 (Actual)

PRIMARY OUTCOMES:
Eyelid margin erythema | Two weeks

SECONDARY OUTCOMES:
Signs and symptoms of Blepharitis | One week, two weeks, three weeks, four weeks

CONTACTS AND LOCATIONS:
Overall Officials: Reza Haque, MD, PhD, Study Chair — Medical Monitor, Inspire
Locations (33):
- United States (33):
  - Jones Eye Institute, Little Rock, Arkansas
  - Sall Medical Research Center, Artesia, California
  - Milton Hom, OD, Azusa, California
  - The Jules Stein Eye Institute UCLA Laser Refractive Center, Los Angeles, California
  - North Valley Eye Medical Group, Mission Hills, California
  - David Wirta, MD, Inc., Newport Beach, California
  - North Bay Eye Associates, Petaluma, California
  - West Coast Eye Care, San Diego, California
  - Wolstan Eye Associates, Torrence, California
  - Eye Center - A Medical and Surgical Group, Hamden, Connecticut
  - Florida Eye Microsurgical Institute, Boynton Beach, Florida
  - Eye Centers of Florida, Fort Myers, Florida
  - NorthShore University HealthSystems, Glenview, Illinois
  - Chicago Cornea Consultants, Hoffman Estates, Illinois
  - Indiana University School of Medicine, Ophthalmology Dept., Indianapolis, Indiana
  - Eye Physicians and Surgeons, LLP, Iowa City, Iowa
  - Koffler Vision Group, Lexington, Kentucky
  - Wilmer Eye Institute, Johns Hopkins Hospital, Baltimore, Maryland
  - Ophthalmic Consultants of Boston, Boston, Massachusetts
  - Minnesota Eye Consultants, Minneapolis, Minnesota
  - Ophthalmology Associates, St Louis, Missouri
  - Ophthalmology Consultants, St Louis, Missouri
  - Brar-Parekh Eye Associates, Woodland Park, New Jersey
  - South Shore Eye Care, Wantagh, New York
  - Mundorf Eye Center, Charlotte, North Carolina
  - TLC Laser Eye Center, Greensboro, North Carolina
  - Cornerstone Eye Care, High Point, North Carolina
  - Abrams Eye Center, Cleveland, Ohio
  - Bucci Laser Vision Institute, Wilkes-Barre, Pennsylvania
  - McCabe Vision Center, Murfreesboro, Tennessee
  - Eye Clinic of Austin, Austin, Texas
  - See Clearly Vision Group, McLean, Virginia
  - Virginia Eye Consultants, Norfolk, Virginia